CLINICAL TRIAL: NCT00003589
Title: Randomized Study With New Combination Chemotherapies in Advanced Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-08975; EORTC-08975
Record Dates: First submitted 1999-11-01; First posted 2004-07-13 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating advanced non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of three different combination chemotherapy regimens in treating patients who have advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall survival between paclitaxel/cisplatin (arm I), gemcitabine/cisplatin (arm II), and paclitaxel/gemcitabine (arm III) in patients with advanced non-small cell lung cancer. II. Determine the response rate, duration of response, progression-free survival, toxicity, and quality of life of these patients randomized in these three treatment arms.

OUTLINE: This is randomized, multicenter study. Patients are stratified according to performance status (0-1 vs 2) and stage of disease (locally advanced vs metastatic). Patients are randomized to receive paclitaxel IV over 3 hours on day 1 followed by cisplatin IV on day 1 every 3 weeks (arm I), gemcitabine IV over 30-60 minutes on days 1 and 8 and cisplatin IV on day 1 every 3 weeks (arm II), or paclitaxel IV over 3 hours on day 1 followed by gemcitabine IV over 30-60 minutes on days 1 and 8 every 3 weeks (arm III). Patients receive at least 2 courses of treatment. In the absence of unacceptable toxicity and disease progression, patients may receive up to 6 courses of treatment. Quality of life is assessed before, during, and at the end of treatment, then every 6 weeks until disease progression, and then every 3 months until death. Patients are followed every 6 weeks until disease progression, then every 3 months until death.

PROJECTED ACCRUAL: A total of 450 patients (150 patients per arm) will be accrued into this study over 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced non-small cell lung cancer that is progressive within 2 months prior to study entry Stage IIIB due to malignant pleural effusion or supraclavicular lymph node involvement only Stage IV At least 1 bidimensionally or unidimensionally measurable target lesion Brain metastases or leptomeningeal disease that have been treated with radiotherapy, is stable without medications (e.g., steroids), and asymptomatic are allowed

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Prothrombin time less than 1.5 times normal Hepatic: Bilirubin no greater than 1.25 times upper limit of normal (ULN) (no greater than 2.5 times ULN if due to liver metastases) AST or ALT less than 3 times ULN (no greater than 5 times ULN if due to liver metastases) Renal: Creatinine clearance at least 60 mL/min Cardiovascular: No uncontrolled cardiac disease, sign of cardiac failure, or rhythm disturbances requiring medication No myocardial infarction in the past 3 months Neurological: No preexisting motor or sensory neurotoxicity of grade 2 or greater Other: No active uncontrolled infection Not a poor medical risk due to nonmalignant disease No secondary primary malignancy in the past 5 years (excluding melanoma, breast cancer, and hypernephroma) except carcinoma in situ of the cervix or adequately treated basal cell carcinoma of the skin No psychological condition that might hamper compliance in this study Not pregnant Effective contraception required of all fertile patients during and for 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy No concurrent colony stimulating factor except for secondary prophylaxis in case of infection and severe neutropenia No concurrent immunotherapy Chemotherapy: No prior chemotherapy for advanced disease, including intracavitary chemotherapy At least 1 year since prior neoadjuvant or adjuvant chemotherapy No concurrent chemotherapy Endocrine therapy: See Disease Characteristics No concurrent hormonal agents (except corticosteroids for antiemetic prophylaxis) Radiotherapy: Prior radiotherapy should not include all target lesions for evaluation At least 4 weeks since prior radiotherapy Concurrent palliative radiotherapy allowed if indicator lesion is outside of radiation field Surgery: Not specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 1998-08; Primary Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Egbert F. Smit, MD, Study Chair — Free University Medical Center
Locations (33):
- Algemeen Ziekenhuis Middelheim, Antwerp, Belgium
- University Hospital Bulovka, Krhanice, Czechia
- National Cancer Institute of Egypt, Cairo, Egypt
- CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy, France
- Thoraxklinik Rohrbach, Heidelberg, Germany
- Hippokration General Hospital of Athens, Athens, Greece
- Ospedale degli Infermi, Biella, Italy
- Netherlands (21):
  - Leyenburg Ziekenhuis, 's-Gravenhage (Den Haag, the Hague)
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Gelre Ziekenhuizen - Lokatie Lukas, Apeldoorn
  - Arnhems Radiotherapeutisch Instituut, Arnhem
  - Ziekenhuis de Baronie, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Ziekenhuis St Jansdal, Harderwijk
  - Elkerliek Ziekenhuis, Helmond
  - Leiden University Medical Center, Leiden
  - Rijnland Ziekenhuis, Leiderdorp
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Sint Antonius Ziekenhuis, Nieuwegein
  - University Medical Center Nijmegen, Nijmegen
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
  - St. Maartens Gasthuis, Venlo
  - Ziekenhuis de Heel, Zaandam
  - Sophia Ziekehuis, Zwolle
- Maritime Hospital, Gdynia, Poland
- Medical Oncology Centre of Rosebank, Johannesburg, South Africa
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Getafe, Madrid
- Ospedale San Giovanni, Bellinzona, Switzerland

REFERENCES:
- [Background] Giaccone G. Gemcitabine plus taxane combinations in non-small cell lung cancer. Semin Oncol. 1999 Feb;26(1 Suppl 4):19-24. PMID 10201517
- [Result] Efficace F, Bottomley A, Smit EF, Lianes P, Legrand C, Debruyne C, Schramel F, Smit HJ, Gaafar R, Biesma B, Manegold C, Coens C, Giaccone G, Van Meerbeeck J; EORTC Lung Cancer Group and Quality of Life Unit. Is a patient's self-reported health-related quality of life a prognostic factor for survival in non-small-cell lung cancer patients? A multivariate analysis of prognostic factors of EORTC study 08975. Ann Oncol. 2006 Nov;17(11):1698-704. doi: 10.1093/annonc/mdl183. Epub 2006 Sep 12. PMID 16968876
- [Result] Smit EF, van Meerbeeck JP, Lianes P, Debruyne C, Legrand C, Schramel F, Smit H, Gaafar R, Biesma B, Manegold C, Neymark N, Giaccone G; European Organization for Research and Treatment of Cancer Lung Cancer Group. Three-arm randomized study of two cisplatin-based regimens and paclitaxel plus gemcitabine in advanced non-small-cell lung cancer: a phase III trial of the European Organization for Research and Treatment of Cancer Lung Cancer Group--EORTC 08975. J Clin Oncol. 2003 Nov 1;21(21):3909-17. doi: 10.1200/JCO.2003.03.195. PMID 14581415